CLINICAL TRIAL: NCT00715234
Title: Evaluation of Vaccination Reminder/Recall Systems for Adolescent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-0763; U01IP000129 (NIH)
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Human Papilloma Virus (HPV); Tetanus-diphtheria-acellular Pertussis (Tdap); Meningococcal Infection; Varicella
Keywords: adolescent reminder/recall; adolescent vaccines; Tdap; Meningococcal; HPV; Reminder cards; Recall messages; vaccine; conjugate
MeSH Terms: conditions — Meningococcal Infections; Chickenpox | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reminder/recall notices for vaccines (Experimental): This group will receive up to 4 recall messages (both letters and computer-generated phone messages) reminding them to get their vaccines. There are 4 separate study groups: 1) private pediatric patients 2) public pediatric patients 3) school-based health center patients and 4) family medicine patients.
  Interventions: Other: Reminder/recall notices for vaccines
- Usual Care (No Intervention): This group will receive usual care. There are 4 separate study groups: 1) private pediatric patients 2) public pediatric patients 3) school-based health center patients and 4) family medicine patients.

INTERVENTIONS:
Other: Reminder/recall notices for vaccines — 1. Receive a generic letter reminding them to make an appointment to get vaccines.
  2. Receive a computer-generated telephone message at 1 week post initial letter.
  3. Receive a computer-generated telephone message at 2 months post initial letter.
  4. Receive a letter at 3 months post initial letter.
  Arms: Reminder/recall notices for vaccines

SUMMARY:
A study team with extensive experience in immunization delivery research will evaluate the effectiveness of vaccination reminder/recall systems for adolescent patients in five types of clinical settings including: urban pediatric, urban family medicine and rural family medicine practices, public pediatric clinics, and school-based health centers. Randomized controlled trials of reminder/recall for adolescents will be conducted at each type of site, with randomization at the level of the patient.

DETAILED DESCRIPTION:
Although patient reminder/recall systems have been shown to be effective at improving vaccination coverage levels for infants and younger children, little is known about the effectiveness of such systems for increasing immunization rates in adolescent populations. The process of reminder/recall in adolescents, and vaccination of adolescents overall, presents particular challenges. Adolescents are less likely to routinely access health care compared to younger children and adults. In addition, other obstacles such as lack of health insurance, missed opportunities for vaccination during health care visits, and the scattering of immunization records across multiple providers have posed major challenges in the vaccination of adolescents. Issues of parental consent for vaccination can also be problematic, given that adolescents may present for care without their parents accompanying them. These and other barriers to immunization may reduce the effectiveness of reminder/recall for adolescents. In the current research study, a study team with extensive experience in immunization delivery research will investigate the ability of pediatricians and family physicians in a number of different practice settings to implement a reminder/recall system for their adolescent patient populations. In addition, we will be able to examine the effectiveness of reminder/recall originating at public school-based health centers, an innovative strategy that has not previously been reported. Randomized controlled trials of reminder/recall for adolescents will be conducted at each type of site. The study team will track important process measures during reminder/recall including the percentage of the eligible population who actually received intervention; percentage with incorrect addresses; percentage with incorrect or disconnected phones; percentage actually up-to-date but incorrectly recalled; missed vaccination opportunities; and invalid doses of vaccines administered. In this way, we will be able to not only determine the degree to which reminder/recall was successful for adolescents, but also identify impediments to success, which will provide a foundation for future efforts. Our study will also investigate the cost of establishing and operating a reminder/recall system for adolescents in each type of clinical setting.

Major Hypotheses

1. Reminder/recall of adolescents will result in an increased rate of receipt of immunizations in private settings of approximately 10 percentage points
2. Reminder/recall will result in a greater rate of receipt of immunizations when patients in public settings have access to a school-based health center (SBHC) compared to when they do not have access to a SBHC
3. Reminder/recall originating at SBHC sites will result in the highest efficacy of reminder/recall among all the types of clinical sites

ELIGIBILITY:
Inclusion Criteria:

* children ages 11-18
* seen in practice in last 2 years
* not up-to-date on any or all shots (Tdap, HPV, meningococcal)
* parents agree to participate in Colorado Immunization and Information System registry

Exclusion Criteria:

* up-to-date on all vaccines
* under age 11 over age 18
* patients who have moved or gone elsewhere at each practice setting

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4807 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
1) the percentage receiving any vaccine after the baseline time point | 6 months after intervention
The percentage of adolescents becoming up-to-date on all needed immunizations | 6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, MPH, Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Background] Ziv A, Boulet JR, Slap GB. Utilization of physician offices by adolescents in the United States. Pediatrics. 1999 Jul;104(1 Pt 1):35-42. doi: 10.1542/peds.104.1.35. PMID 10390257
- [Background] Schaffer SJ, Humiston SG, Shone LP, Averhoff FM, Szilagyi PG. Adolescent immunization practices: a national survey of US physicians. Arch Pediatr Adolesc Med. 2001 May;155(5):566-71. doi: 10.1001/archpedi.155.5.566. PMID 11343499
- [Background] Briss PA, Rodewald LE, Hinman AR, Shefer AM, Strikas RA, Bernier RR, Carande-Kulis VG, Yusuf HR, Ndiaye SM, Williams SM. Reviews of evidence regarding interventions to improve vaccination coverage in children, adolescents, and adults. The Task Force on Community Preventive Services. Am J Prev Med. 2000 Jan;18(1 Suppl):97-140. doi: 10.1016/s0749-3797(99)00118-x. PMID 10806982
- [Background] Humiston SG, Rosenthal SL. Challenges to vaccinating adolescents: vaccine implementation issues. Pediatr Infect Dis J. 2005 Jun;24(6 Suppl):S134-40. doi: 10.1097/01.inf.0000166161.12087.94. PMID 15931141
- [Background] Szilagyi PG, Bordley C, Vann JC, Chelminski A, Kraus RM, Margolis PA, Rodewald LE. Effect of patient reminder/recall interventions on immunization rates: A review. JAMA. 2000 Oct 11;284(14):1820-7. doi: 10.1001/jama.284.14.1820. PMID 11025835
- [Background] Kempe A, Lowery NE, Pearson KA, Renfrew BL, Jones JS, Steiner JF, Berman S. Immunization recall: effectiveness and barriers to success in an urban teaching clinic. J Pediatr. 2001 Nov;139(5):630-5. doi: 10.1067/mpd.2001.117069. PMID 11713438
- [Derived] Suh CA, Saville A, Daley MF, Glazner JE, Barrow J, Stokley S, Dong F, Beaty B, Dickinson LM, Kempe A. Effectiveness and net cost of reminder/recall for adolescent immunizations. Pediatrics. 2012 Jun;129(6):e1437-45. doi: 10.1542/peds.2011-1714. Epub 2012 May 7. PMID 22566415